CLINICAL TRIAL: NCT01646697
Title: Cytopathologic Margin Evaluation in Patients Undergoing Pancreatic Cancer Resection
Brief Title: Slide Interpretation or Standard Surgical Pathology in Assessing Margin Status in Patients With Pancreatic Cancer Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-10110; NCI-2012-00926 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Pancreatic Cancer; Adenocarcinoma
Keywords: pancreatic cancer; adenocarcinoma; pancreatic resection
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (cytopathologic evaluation) (Experimental): Patients undergo cytopathologic sample collection during pancreatic resection during which slides are gently pressed against the cut edge of the pancreas, the surgical bed, and along the superior mesenteric artery, and finally against the tumor itself.
  Interventions: Other: cytology specimen collection procedure

INTERVENTIONS:
Other: cytology specimen collection procedure — Undergo cytopathologic sample collection
  Other Names: cytologic sampling

SUMMARY:
This study is being done to investigate another way of evaluating margin status after pancreatectomy by using cytopathology (slide interpretation) as compared to the traditional method of surgical pathology

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare margin status on final pathology with margin status from cytopathologic evaluation.

OUTLINE:

Patients undergo cytopathologic sample collection during pancreatic resection during which slides are gently pressed against the cut edge of the pancreas, the surgical bed, and along the superior mesenteric artery, and finally against the tumor itself.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing pancreatic resection for a presumed, although not necessarily biopsy-proven pancreatic malignancy,
* ages 18 years to 80 years old

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-11-07 (Actual); Primary Completion 2016-02-06 (Actual); Study Completion 2016-02-06 (Actual)

PRIMARY OUTCOMES:
Local recurrence at the site of resection | up to 2 years
  Will be evaluated in a Cox proportion hazards regression model. The prognostic ability of the histological reporting of the specimen margin as well as the cytopathological reporting of the specimen and in situ margins will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bloomston, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu